CLINICAL TRIAL: NCT00639275
Title: Effects of Subthalamic Nucleus Deep Brain Stimulation on Gastrointestinal Symptoms and Motility in Parkinson's Disease.
Brief Title: Deep Brain Stimulation and Digestive Symptomatology
Acronym: SCPDig
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/050/HP
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with Parkinson's disease (PD) frequently experience upper gastrointestinal disorders. During the disease, weight loss is often noticed. Recently, many studies have demonstrated that STN-DBS improved extrapyramidal symptoms. Interestingly, PD patients gain weight after STN-DBS, at least in part due to a decrease in resting energy expenditure.

Purpose: To evaluate benefits of STN-DBS on upper gastrointestinal symptoms and motility.

Patients et method: PD patients waiting for STN-DBS, will be assessed in a preoperative time (2 times at, at least, 3 month intervals, to evaluate the natural history of the disease on upper gastrointestinal symptoms and motility) and in a postoperative time, after 6 months of chronic STN-DBS. Each assessment will include : 1/ questionnaires about frequency and severity of upper gastrointestinal symptoms; 2/ a nutritional assessment (body mass index, dietary assessment); 3/ the gastric emptying measurement with the 13C-octanoic acid breath test; 4/ the colorectal transit time measurement with radio-opaque markers 5/ an indirect calorimetry to estimate resting energy expenditure; 6/ and plasmatic leptin and ghrelin concentrations, hormones involved in the homeostatic regulation of appetite.

Perspectives: This physiopathological study should allow us to understand the mechanisms of the effects of STN-DBS on upper gastrointestinal symptoms and weight regulation in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Electrode implantation for deep brain stimulation in progress
* Age <70 yr
* Motor fluctuations and dyskinesias
* Motor symptoms improvement with L-dopa > 50%
* No dementia
* No depression
* No major psychiatric symptom
* Normal brain MRI

Exclusion Criteria:

* Contra-indication of neurosurgery
* Pregnancy
* Diabetes
* Obesity
* Compulsive eating disorders
* Organic digestive disease
* Gastrointestinal resection
* Prokinetic treatment
* Coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients with subthalamic nucleus deep brain stimulation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
the gastric emptying measurement with the 13C-octanoic acid breath test | M0 and M6

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France